CLINICAL TRIAL: NCT02593383
Title: A Placebo Control, Multicenter, Randomized, Double Blind, Multi-formula Groups, and Parallel Phase Ⅰb+Ⅱa Study Evaluating the Safety and Efficacy of Compound Adapalene and Clindamycin Hydrochloride Gel in Treatment of Patients With Acne
Brief Title: Compound Adapalene and Clindamycin Hydrochloride Gel in Treatment of Patients With Acne
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: zhaoke-2015-02
Record Dates: First submitted 2015-07-16; First posted 2015-11-02 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Acne
Keywords: safety; efficacy
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Clindamycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Treat group 1 (Experimental): Group 1: 0.1% Adapalene + 1% Clindamycin Hydrochloride
  Interventions: Drug: Adapalene + Clindamycin Hydrochloride
- Treatment group 2 (Experimental): Group 2: 0.1% Adapalene + 2% Clindamycin Hydrochloride
  Interventions: Drug: Adapalene + Clindamycin Hydrochloride
- Treatment group 3 (Experimental): Group 3: 0.05% Adapalene + 0.5% Clindamycin Hydrochloride
  Interventions: Drug: Adapalene + Clindamycin Hydrochloride
- Treatment group 4 (Experimental): Group 4: 0.05% Adapalene + 1% Clindamycin Hydrochloride
  Interventions: Drug: Adapalene + Clindamycin Hydrochloride
- Placebo group (Placebo Comparator): Placebo Group: Blank Gel
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adapalene + Clindamycin Hydrochloride — 0.1% Adapalene + 1% Clindamycin Hydrochloride
  Arms: Treat group 1
Drug: Adapalene + Clindamycin Hydrochloride — 0.1% Adapalene + 2% Clindamycin Hydrochloride
  Arms: Treatment group 2
Drug: Adapalene + Clindamycin Hydrochloride — 0.05% Adapalene + 0.5% Clindamycin Hydrochloride
  Arms: Treatment group 3
Drug: Adapalene + Clindamycin Hydrochloride — 0.05% Adapalene + 1% Clindamycin Hydrochloride
  Arms: Treatment group 4
Drug: Placebo
  Arms: Placebo group

SUMMARY:
evaluate the safety and efficacy of Compound Adapalene and Clindamycin Hydrochloride Gel in treatment of chinese patients with acne.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 40 years old, female or male;
2. Class I-III of Acne vulgaris according to the International Modified PILLSBURY Classification;
3. Patients voluntarily take part in the study and sign the ICF.

Exclusion Criteria:

1. The subject is known to be allergic to adapalene, clindamycin hydrochloride, clindamycin, and / or any components of gel excipient;
2. Patients with secondary acne including occupational acne and corticosteroid-induced acne;
3. The affected skin has other concomitant lesion (such as solar dermatitis, psoriasis, seborrheic dermatitis, eczema and extremely severe acne) which may impact the efficacy evaluation;
4. Subject has the history of regional enteritis, ulcerative colitis or antibiotic-associated colitis;
5. Patient has history of severe cardiac disease and hypertension;
6. Patient has severe liver and kidney diseases with AST/ALT more than twice upper limitation, or Cr, total cholesterol and triglycerides above normal range;
7. Patients with severe endocrine diseases, blood diseases, and neuropsychiatric disorders;
8. Patients are known to have severe immune dysfunction, or need long-term use of corticosteroids or immunosuppressive agents;
9. Pregnant or breastfeeding women, or unwilling to take effective contraceptive measures during the study;
10. Alcoholic patients or drug abusers;
11. Patient has used other acne drugs topically within 2 weeks before the study start;
12. Patient has been administered with victoria A acid, vitamins, and antibiotics within 4 weeks before the study start;
13. Patient has participated in other study within 3 months before the study start;
14. The subject is not fit to take part in this study in the judgment of the investigator.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 245 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
efficacy endpoint | 12 weeks
  number of patients with deceased acne lesions at the treatment end (Day 85±3) in each group;

SECONDARY OUTCOMES:
IGA classification change | 12 weeks
  The improvement of IGA （investigator general Assess）Classification at the treatment end (Day 85±3) in each group
treatment success rate | 12 weeks
  The treatment success rate at the treatment end (Day 85±3) in each group; calculation methods:number of patients with IGA assessment improved to level 0 to level 1/ total number of patients
PK | 12 weeks
  AUC
PK | 12 weeks
  peak plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Heng GU, MD, Principal Investigator — Institute of Dermatology, Chinese Academy of Medical Sciences
Locations (1):
- Institute of Dermatology, Chinese Academy of Medical Sciences, Nanjing, Jiangsu, China